CLINICAL TRIAL: NCT01223963
Title: A Multi-center Retrospective Chart Review of Medical Records on the Use of Macrolane Volume Restoration Factor for Breast Enhancement
Brief Title: Macrolane Retrospective Study
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: 31GB0902
Record Dates: First submitted 2010-10-15; First posted 2010-10-19 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2012-11

CONDITIONS: Women Who Have Had Breast Enhancement With Macrolane VRF
Keywords: Macrolane; Retrospective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Macrolane: Women that have had breast enhancement with Macrolane Volume Restoration Factor.

SUMMARY:
This is a retrospective, multicenter chart review of medical records on the use of Macrolane for female breast enhancement.

The primary objective is to evaluate the safety profile of Macrolane Volume Restoration Factor 20 and Macrolane Volume Restoration Factor 30 when used for female breast enhancement in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Females treated with Macrolane Volume Restoration Factor 20 and/or Volume Restoration Factor 30 for breast enhancement.
* Signed Informed Consent

Exclusion Criteria:

* Subjects that have actively asked not to be contacted by the clinic
* Subjects that have participated or participates in clinical studies with Macrolane for breast enhancement

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women that have had breast enhancement in clinics in Sweden (and UK).
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, Md PhD, Principal Investigator — Akademikliniken
Locations (4):
- Sweden (4):
  - Stureplanskliniken, Gothenburg
  - Akademikliniken, Malmo
  - Stureplanskliniken, Stockholm
  - Akademikliniken, Stockholm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Macrolane
Started | 93 (All subjects treated between May 1 2008 and Dec 31 2009 in selected clinics were to be asked.)
Completed | 93
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Macrolane
Number analyzed (Participants) | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 93
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Number of Adverse events reported during the study period
Time Frame: 01may2008 - 31dec2009
Measure: Number; unit: number of AE
Groups:
- Macrolane: Number of related Adverse events reported during the study period
Arm/Group | Macrolane
Number analyzed (Participants) | 93
number of AE | 46

2. Other Pre Specified Outcome: Number of Participants Who Reported Being at Least Somewhat Satisfied at Any Tine Post-procedure
Description: The alternative outcomes were: still satisfied, never satisfied, 3-5 months, 6-8 months, 9-11 months, 12 months or more, still satisfied when retreated.
Time Frame: up to 12 months post-procedure
Measure: Number; unit: participants
Arm/Group | Macrolane
Number analyzed (Participants) | 93
participants | 89

ADVERSE EVENTS:
Arm/Group | Macrolane
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 21/93
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macrolane (N=93)
Capsular contracture associated with breast implant (General disorders) | 21
Implant site nodule (General disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less